CLINICAL TRIAL: NCT06187389
Title: Assessing the Validity and Reliability of the Turkish Version of the 4AT Scale in Post-Anesthesia Awakening Delirium
Brief Title: Validation and Reliability of the Turkish 4AT Scale for Post-Anesthesia Awakening Delirium
Status: Completed | Type: Observational
Sponsor: Kilis 7 Aralik University (Other)
Responsible Party: Principal Investigator, İslam Elagöz, Principal Investigator, Kilis 7 Aralik University
Other Study IDs: kilis7aralıkU1
Record Dates: First submitted 2023-12-16; First posted 2024-01-02 (Actual); Last update posted 2024-01-02 (Actual); Status verified 2023-12

CONDITIONS: Delirium; Awakening, Post-Anesthesia Delayed; Delirium, Postoperative; Nurse's Role; Nursing Caries
MeSH Terms: conditions — Delirium; Delayed Emergence from Anesthesia; Emergence Delirium

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: 1 Grups — This methodological study was conducted using a cross-sectional observational approach at a leading teaching and research hospital. The study duration was from March to June 2023

SUMMARY:
Background: Delirium is a common and serious condition in hospitalized patients that often leads to extended hospital stays and increased healthcare costs. Accurate and timely detection is essential for optimal patient outcome.

Aims: This study aimed to adapt the internationally recognized 4 AT Delirium Diagnosis Scale to Turkish and to evaluate the validity and reliability of this tool for the Turkish patient population.

Design: This study was structured and conducted at a state hospital from March to June 2023.

Methods: The study included 188 participants, determined through a power analysis. The 4AT Delirium Test and additional assessment tools were used to ascertain the delirium status of the patients. Comprehensive statistical evaluations were conducted using SPSS 25.0, which included analyses, such as item difficulty indices, item discrimination, and chi-square tests. Ethical approval for this study was granted by the Non-Interventional Ethics Committee, ensured full compliance with the ethical standards set by the World Medical Association's Declaration of Helsinki. All participants provided informed consent before participation. Additionally, our results strictly adhered to the guidelines of the STROBE Checklist.

DETAILED DESCRIPTION:
Delirium is a common occurrence in healthcare settings, leading to extended hospital and intensive care stays, and negatively impacting mortality and morbidity rates [1,2]. Previously seen as an unavoidable outcome, delirium is now understood as a preventable condition [3,4]. The delirium incidence in postoperative recovery units fluctuates between 3% and 54%, contingent upon the diagnostic method, patient demographics, and timing of the assessment [6,7,8,9].

Although a myriad of approaches and scales are employed to detect delirium, some may inadequately or erroneously define the condition. Overlooking delirium in its early stages increases healthcare expenses, extends hospitalization, burdens healthcare staff, and interrupts therapeutic plans [3,10,11]. Additionally, the importance of credible and efficient evaluation methods for delirium detection in postoperative recovery units has been underscored [6]. Both the Anesthesia Association and the European Anesthesia Association emphasize the significance of early delirium identification in these units [12,13]. Delirium onset in recovery units correlates with its emergence in general wards or intensive care units [14]. Thus, patients should not be discharged from the recovery units without undergoing a delirium assessment.

A comprehensive psychiatric evaluation remains a benchmark for diagnosing delirium. However, given the extensive training this method demands and its lengthy process [15,16] , there is a need for more streamlined and promptly applicable tests for routine delirium screening in postoperative recovery units. While many scales used for delirium assessment require specialized training and are time intensive [17,18], tools such as the delirium risk determination scale, confusion assessment method [CAM] [19], confusion assessment scale for the ICU [CAM-ICU] [20], 3D confusion assessment method [3D-CAM], delirium index [DI], and confusion assessment method importance [CAM-S] have gained acceptance. However, many of these tools are unwieldy [9,17,18]. In response, the 4 At Delirium screening scale [4 AT] was formulated for more rapid and dependable delirium screening [21,22].

The 4AT is a concise assessment tool, comprised of four items designed to evaluate delirium. Healthcare professionals can administer this test in less than 2 minutes, eliminating the need for specialized training [21]. The efficacy of 4AT has been validated in numerous studies involving various populations [21,23,24]. Despite its global recognition and adoption as a clinical instrument, there is a noticeable gap in research on its application within postoperative recovery units, or "awakening units," using the 4AT scale.

Screening for delirium, particularly following surgery, is crucial for timely identification because of its significant impact on long-term patient outcomes. Thus, there is an undeniable demand for reliable and streamlined assessment instruments. Many current tools require specialized knowledge and can be unwieldy in applications. A notable gap exists within Turkey's postoperative recovery setting for efficient and trustworthy delirium screening methods. Against this backdrop, our research aims to tailor the internationally recognized 4 AT Delirium Diagnosis Scale to the Turkish landscape and confirm its effectiveness. The primary objective of this study was to adapt the 4 AT Delirium Diagnosis Scale for Turkish use and ascertain its validity and reliability in a Turkish patient cohort. Within this framework, we address the following questions.

1. What is the validity of the 4 AT Delirium Test for the Turkish patient population?
2. What is the reliability of the 4 AT Delirium Test for the Turkish patient population?

ELIGIBILITY:
Inclusion Criteria:

* Our study cohort comprised patients who satisfied certain prerequisites. These included being aged 18 years or older, possessing the capability to communicate, scoring between -3 and +4 on the Richmond Agitation-Sedation Scale [RASS], achieving a minimum score of 10 on the Glasgow Coma Scale [GCS], and no neurological or psychiatric backdrop that might skew a delirium assessment. If any participant opted to exit the study, their associated data were omitted.

Exclusion Criteria:

* Individuals who encountered acute post-anesthesia complications, were diagnosed with advanced cognitive deficits or dementia, lost communication abilities entirely, or displayed reluctance or inability to furnish information during the study were excluded. Moreover, patients diagnosed with an alternate neurological or psychiatric ailment after delirium assessment were also included. Participants or their guardians, who either declined involvement or retracted prior consent, were excluded from the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The study population consists of adult patients admitted to the ICU for surgery. Participants were selected based on preoperative cognitive status assessments, with those showing normal evaluations included in the study. The population exhibits diversity in terms of age, gender, and types of surgery. Post-operative patients in the recovery room were evaluated for consciousness and sedation agitation levels using established scales such as RASS and GKS. The study specifically focuses on screening for post-anesthesia emergence delirium, making the population representative of typical ICU surgical cases where delirium assessment is critical
Sampling Method: Non-Probability Sample
Enrollment: 188 (Actual)
Dates: Start 2023-03-01 (Actual); Primary Completion 2023-05-01 (Actual); Study Completion 2023-06-01 (Actual)

PRIMARY OUTCOMES:
Patient evaluation form: The patient Evaluation Form | up to 12 weeks
  Crafted by the research team to delve into potential delirium triggers and capture anamnestic information gathered during the patient's initial check-in. Beyond capturing basic demographics such as age, sex, marital status, and education, the form delves deep into the patient's overall health profile, lifestyle, and associated risk factors.
Richmond Sedation-Agitation Scale [RASS]: | up to 12 weeks
  This scale offers a thorough observational evaluation. Initially, the patient's sedative status was gauged. If the patient is profoundly sedated, unresponsive, or registers a score between -4 and -5 on the RASS, no assessment can be performed. In these deep sedative states, often termed comas or stupors, the patient does not react to stimuli, rendering delirium evaluation moot. However, as soon as patients become alert [RASS> -3], delirium assessments are feasible. The scale operates on a scoring system ranging from +4 to -5.
The Glasgow Coma Scale [GCS], | up to 12 weeks
  which is globally recognized and adopted in ICUs, was conceived by Teasdale and Jennet in 1974 to exclusively gauge consciousness levels in patients with traumatic brain injury. This scale delineates separate evaluation criteria for the adult and pediatric cohorts. Rooted in three core categories, GCS is a physiological scoring mechanism to monitor patients' clinical trajectory from admission throughout their hospital tenure. Only patients with a GCS score ≥ 10 were deemed suitable for delirium evaluation
Confusion Assessment Metot in the Intensive Care Unit [Cam-ICU]: | up to 12 weeks
  Tailored for ICU-based confusion assessments, the Cam-ICU operates on DSM-V parameters and is completed in under five minutes
Nursing Delirium Screening Scale [Nu-DESC] | up to 12 weeks
  The Nu-DESC is a 5-item observational tool geared towards rapid delirium detection. The scale encompasses elements, such as disorientation, inappropriate conduct, flawed communication, hallucinations, and psychomotor retardation. Each facet was scored between 0 and 2, with aggregate scores capped at 10. Individuals with scores of ≥ 2 were labeled as delirious.
4AT Delirium Test: | up to 12 weeks
  The Turkish adaptation of the 4AT was curated in alignment with the guidelines delineating the cross-cultural adaptation of health-centric scales. Under the guidance of the original creator, Prof. Alasdair M.J. MacLullich from the University of Edinburgh translated the Turkish 4AT by a trio comprising two English academics and a psychiatrist. The subsequent phase entailed bilingual academic nurses unfamiliar with the 4AT, executing a back-translation. After test-driving the translation on assorted samples, the final version was greenlit for the 4AT application. The 4AT, a user-friendly delirium and cognitive disorder assessment tool, is a breeze for practitioners to administer and does not require specialized training.

CONTACTS AND LOCATIONS:
Overall Officials: islam elagöz, MsC, Study Chair — kils 7 aralık University
Locations (1):
- Islam Elagöz, Kilis, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
"In this study, we do not plan to share individual participant data with other researchers. The decision not to share IPD is based on concerns related to participant privacy and confidentiality. The data collected in this study are sensitive and disclosing them, even in a de-identified format, could pose risks to participant privacy. Therefore, in accordance with our ethical obligations and institutional guidelines, we have decided to maintain the confidentiality of the data and not make it available for external access.